CLINICAL TRIAL: NCT04734899
Title: The Effects of Foot-Core Training on Muscle Activations, Walking, Balance and Lower Extremity Performance in Individuals With Pes Planus
Brief Title: Foot Core Training in Individuals With Pes Planus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Assistant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/15-04
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pes Planus
Keywords: Pes planus; Electromyography; Gait; Balance
MeSH Terms: conditions — Flatfoot | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial: Two parallel treatment groups; The control group will only receive exercise therapy, while the other group will receive foot core training in addition to exercise therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control grup (Active Comparator): All individuals participating in the study will be taught the exercises given to strengthen weakened muscles, stretch shortened structures and increase proprioception by the physiotherapist and will be asked to do these exercises at least twice a day for 8 weeks.
  The home program will be followed by the exercise daily form.
  Interventions: Other: Exercise program
- Foot core grup (Experimental): In addition to the exercise program given to the control group, foot core training will be added and taught by the physiotherapist and they will be asked to do these exercises at least twice a day for 8 weeks.
  Interventions: Other: Exercise program; Other: Foot core training

INTERVENTIONS:
Other: Exercise program — Strengthening with resistance bands for tibialis posterior, tibialis anterior, peroneus longus, finger flexors, hip and knee muscles, sheet gathering exercises, fingertip walking exercises, Stretching exercises for gastrocnemius and soleus muscles, plantar fascia stretching, weight transfer on one leg
Other: Foot core training — Short foot exercises with passive modeling, active assisted modeling, active modeling, functional training
  Arms: Foot core grup

SUMMARY:
Foot core training is very important for the intrinsic muscles of the foot, but it is often neglected in exercise programs given to individuals with pes planus. The aim of our study is to reveal the effects of foot core training, which will be added to the exercise program routinely given to individuals with asymptomatic flexible pes planus, on walking, muscular activations, balance and lower extremity functional performance with objective, evidence based results.

DETAILED DESCRIPTION:
This study is a randomized controlled study and will be carried out on volunteer individuals with asymptomatic flexible pes planus aged between 18-25, studying at Alanya Alaaddin Keykubat University. Persons meeting the inclusion criteria will be determined by the specialist physiotherapist. Surface electromyography (sEMG) measurements will be made by a doctorate physiotherapist. Other evaluations will be made by a specialist physiotherapist. Individuals who meet the inclusion criteria, who volunteered to participate in the study and signed the consent sheet will be randomly divided into two groups, the control group and the foot core group. Individuals with initial evaluations will be followed up in an exercise program planned for 8 weeks. The control group will be given exercises to strengthen the weakened muscles, stretch the shortened structures and increase proprioception. Foot core training will be given to the study group in addition to the exercises given to the control group. Before and after exercise, the subjects will be assessed with navicular height measurement, muscle activation evaluation, evaluation of walking parameters, functional lower extremity performance evaluation and balance evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteer to participate in the study
* Individuals between the ages of 18-25
* Individuals with a body mass index between 18.5-30.
* Individuals with a difference of 10 mm or more between weighted and unweighted measurements by applying the navicular drop test
* Individuals who are considered to have flexible pes planus with a positive Jack's finger lift test

Exclusion Criteria:

* Individuals with symptoms such as any pain in the foot and ankle, fatigue.
* Individuals with any neurological or orthopedic disease affecting the lower extremity.
* Individuals with a history of foot-ankle trauma-surgery
* Individuals with lower extremity inequality of more than 1 centimeter (cm)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of muscle activation | Change from baseline muscle activation at 8 weeks
  In our study, muscle activations of the tibialis anterior, peroneus longus and abductor hallucis muscles both during maximum isometric contraction and during walking will be evaluated by a trained and experienced researcher using the sEMG device.

SECONDARY OUTCOMES:
Y balance test (YBT): | Just before the training and at the end of 8-week training
  There are 3 bars of 1.5 meters long fixed to a 2.54 cm high central foot plate at an angle of 135 and 90 degrees between them. It is asked to lie down with the tip of the toe in 3 directions and the measurements are recorded.
Vertical jump, flight time | Just before the training and at the end of 8-week training
  Vertical jumping and jumping on one foot will be evaluated with MicroGate Opto-jump Next®. With this test, flight time will be measured during vertical jump, and it will be recorded by seconds.
Vertical jump, jump height | Just before the training and at the end of 8-week training
  Vertical jumping and jumping on one foot will be evaluated with MicroGate Opto-jump Next®. Jump height wil be recorded by centimeters.
Vertical jump, power | Just before the training and at the end of 8-week training
  Vertical jumping and jumping on one foot will be evaluated with MicroGate Opto-jump Next®. Power will be recorded by watt/kilogram.
vertical jump, position difference | Just before the training and at the end of 8-week training
  Vertical jumping and jumping on one foot will be evaluated with MicroGate Opto-jump Next®. Position difference will be measured by centimeters.
Cadence | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and as a result of the analysis cadence will be recorded as steps per minute.
Gait speed | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and as a result of the analysis, gait speed will be measured as meter/seconds.
Step width | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and step width will be measured as centimeter.
Ratio of step length to step height | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and as a result of the analysis, ratio of step length to step height will be calculated as a percentage.
Standing phase duration | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track. Standing phase duration will be recorded as seconds.
Swing phase duration | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track. Swing phase duration will be recorded as seconds.
Double support period duration | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and as a result of the analysis, double support period duration will be recorded as seconds.
Single support period time | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and as a result of the analysis, single support period time will be recorded as seconds.
Acceleration | Just before the training and at the end of 8-week training
  It will be evaluated using a digital miniature gait analysis system. Participants will be asked to walk on the 20-meter track and as a result of the analysis, at what moments and at what speed the acceleration during walking will be reached as seconds and meter/second, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung DY, Koh EK, Kwon OY. Effect of foot orthoses and short-foot exercise on the cross-sectional area of the abductor hallucis muscle in subjects with pes planus: a randomized controlled trial. J Back Musculoskelet Rehabil. 2011;24(4):225-31. doi: 10.3233/BMR-2011-0299. PMID 22142711
- [Background] McKeon PO, Hertel J, Bramble D, Davis I. The foot core system: a new paradigm for understanding intrinsic foot muscle function. Br J Sports Med. 2015 Mar;49(5):290. doi: 10.1136/bjsports-2013-092690. Epub 2014 Mar 21. PMID 24659509
- [Background] Mulligan EP, Cook PG. Effect of plantar intrinsic muscle training on medial longitudinal arch morphology and dynamic function. Man Ther. 2013 Oct;18(5):425-30. doi: 10.1016/j.math.2013.02.007. Epub 2013 Apr 28. PMID 23632367
- [Background] Kim EK, Kim JS. The effects of short foot exercises and arch support insoles on improvement in the medial longitudinal arch and dynamic balance of flexible flatfoot patients. J Phys Ther Sci. 2016 Nov;28(11):3136-3139. doi: 10.1589/jpts.28.3136. Epub 2016 Nov 29. PMID 27942135
- [Background] Glatthorn JF, Gouge S, Nussbaumer S, Stauffacher S, Impellizzeri FM, Maffiuletti NA. Validity and reliability of Optojump photoelectric cells for estimating vertical jump height. J Strength Cond Res. 2011 Feb;25(2):556-60. doi: 10.1519/JSC.0b013e3181ccb18d. PMID 20647944